CLINICAL TRIAL: NCT03948919
Title: Fecal Transplant for Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GI-2019-27285
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FMT Treatment (Active Comparator): Fecal microbiota - 1.0-3.0 x 10^11 CFU / day (2 capsules per day for 8 weeks).
  Interventions: Drug: Fecal microbiota
- Placebo (Placebo Comparator): The placebo consists of a mixture of trehalose and crystalline methylcellulose (Avicel) in 6:1 (w/w) ratio that is packaged in size 0 swedish orange capsules, which are then double encapsulated in size 00 natural colored capsules to make them visibly indistinguishable from encapsulated active product. Two capsules taken daily for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fecal microbiota — Lyophilized encapsulated fecal microbiota given daily for 8 weeks.
  Arms: FMT Treatment
Drug: Placebo — Placebo capsules identical in appearance to fecal microbiota capsules to be taken daily for 8 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the engraftment of donor microbiota with active ulcerative colitis (UC) following sequential fecal microbiota transplant (FMT). One key group of bacteria we are following are sulfate reducing bacteria (SRB). We plan to measure the relative abundance of SRB at baseline and after FMT. It is widely unknown if the microbiota in UC is dysfunctional and therefore perpetuates inflammation, or if the ongoing inflammation shapes the microbiota. We aim to determine if we can alter the microbiota in UC towards a healthy, more diverse microbiota resembling the donor using capsule FMT material.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic, relapsing remitting inflammatory disease of the intestine. The two main forms of IBD are Crohn's disease (CD) and Ulcerative Colitis (UC). There is no cure for IBD and the etiology is unknown, however IBD is thought to arise as an aberrant immune response to the intestinal microbiota. The intestinal microbiota closely correlates with inflammation in IBD. Currently, the treatment of IBD is based on suppressing the aberrant immune response in the intestine. This often takes the form of systemic immunosuppression, which in turn carries a multitude of risks including infection and malignancy. Thus there is an urgent need for safe, effective therapies that ultimately have the potential to cure IBD.

Fecal microbiota transplantation (FMT) is the process of transferring fecal microbiota from one individual to another. FMT has revolutionized the treatment of multiple recurrent Clostridium difficile infection with a cure rate around 90%. Given the success of FMT in C. difficile colitis, attention turned to other forms of colitis, in particular IBD. Early pilot studies demonstrated a mixed result for the use of FMT in IBD. One of the key issues surrounding the use of FMT in IBD is the challenge of engrafting a new microbiota. Additionally IBD flares following FMT for C. difficile infection have been reported, although it is difficult to account for the confounding of the underlying C. difficile infection. This study will examine how FMT donor selection can impact the engraftment of the microbiota into patients with UC.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide consent
* English speaking
* Diagnosis of ulcerative colitis based on typical clinical-histopathic diagnosis
* Diagnosis of ulcerative colitis > 3 months
* Active disease on endoscopy (endoscopic Mayo subscore ≥ 1)
* Evidence of inflammation extending beyond a minimum of 20cm
* Any ongoing ulcerative colitis therapy must be at stable doses for 4 weeks prior to study and remain stable over the course of the study

Exclusion Criteria:

* Extensive bowel resection
* Presence of ileostomy or colostomy
* Suspicion of ischemic colitis, radiation colitis or microscopic colitis
* Diagnosis of Crohn's disease
* Diagnosis of per-anal fistula or abscess
* Adenomatous polyps that have not been removed
* Use of pre or probiotics within 30 days of randomization
* Pregnancy
* Severe food allergies
* End stage liver disease or cirrhosis
* An absolute neutrophil count < 500 cell/µL
* Life expectancy < 6 months

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Engraftment of donor microbiota | 12 weeks
  Engraftment measured by SourceTracker at baseline to week 12 between FMT arm and placebo arm.

SECONDARY OUTCOMES:
Clinical efficacy of FMT versus placebo | 8 weeks
  Change in partial Mayo score from baseline to week 8 between FMT and placebo arm
Clinical efficacy of low sulfate reducing microbiota | 12 weeks
  Partial mayo score at week 12 between those with low sulfate reducing microbiota or not low sulfate reducing microbiota
Rate of change of sulfate reducing microbiota | 4 weeks
  Change in quantitative PCR of sulfate reducing genes at week 1, 2, 3 and 4 between FMT arm and placebo arm
Serious adverse events | 12 weeks
  Number of serious adverse events between FMT arm and placebo arm

CONTACTS AND LOCATIONS:
Overall Officials: Byron Vaughn, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

DOCUMENTS (1):
  • Informed Consent Form (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT03948919/ICF_000.pdf